CLINICAL TRIAL: NCT07077642
Title: Validation of a Multidimensional Scale for the Detection of Health Needs in People With HIV
Acronym: MUSA
Status: Enrolling by invitation | Type: Observational
Sponsor: Giovanni Di Perri (Other)
Responsible Party: Sponsor-Investigator, Giovanni Di Perri, Prof., University of Turin, Italy
Organization: University of Turin, Italy (Other)
Other Study IDs: MUSA
Record Dates: First submitted 2025-06-20; First posted 2025-07-22 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: HIV; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The primary objective is to evaluate the diagnostic performance of the multidimensional screening test in identifying alterations in the domains considered in people with HIV, in order to improve the predictivity of disorders, ensure better care and consequently improve the quality of life of people with HIV

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older

  * Confirmed HIV infection
  * Good understanding of the Italian language
  * Signature of informed consent
  * Inclusion of at least 33% women and at least 33% people older than 50 years of age

Exclusion Criteria:

* Acute ongoing diseases that, in the opinion of the investigators, may affect the performance of the tests (bacterial or viral infections, neoplasms under active chemotherapy treatment)

  * Dementia or other severe neurodegenerative/neurocognitive disorders.
  * Individuals unable to express consent independently and/or supported by protective legal figures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the diagnostic performance of multidimensional screening test in identifying alterations in considered domains in patients with hiv | At enrollment
  Composite endpolint for each domani:
  1. Cognitive impairment (using the Brief Neurocognitive Screening Test)
  2. Depressive symptoms (using the Patient Health Questionnaire-9)
  3. anxiety symptoms (using the General Anxiety Disorder-7 test)
  4. sleep quality (using the Pittsburgh Sleep Quality Index)
  5. quality of life (using the EQ-5D-5L)
  6. functional test (using the Advanced Instrumental Activities of Daily Living Scale)
  7. nutritional (using the Mini Nutritional Assessment (MNA) - short form)
  8. socio-economic (using detailed questions)
  9. stigma (using HIV Stigma Scale - 12 item version, Karolinska Institute)
  10. comorbidities (checking in the medical records)
  11. polytherapy (checking in the medical records)
  12. alcool or drug use (using Audit-C and Brief Substance Craving Scale)

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (11):
  - Università degli Studi di Genova, Genova, Genova
  - ASST Fatebenefratell - Sacco, Ospedale L. Sacco, Milan, Milano
  - Clinica delle Malattie Infettive e Tropicali, Dipartimento di Scienze della Salute, Università degli Studi di Milano, ASST Santi Paolo e Carlo, Milan, Milano
  - Unità di Malattie Infettive, IRCCS San Raffaele, Milan, Milano
  - Ospedale Amedeo di Savoia, Torino, Torino
  - UOC Malattie Infettive, Università di Bari "Aldo Moro", AOU Policlinico di Bari, Bari
  - UOC Malattie Infettive, Arnas Garibaldi, Catania
  - Malattie Infettive ed Urgenze Infettivologiche, Presidio Ospedaliero Cotugno - Azienda Ospedaliera dei Colli, Napoli, Napoli
  - UOC Malattie Infettive e Tropicali, Azienda Ospedale Università di Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS Roma, Roma
  - SS Immunodeficienza, Azienda Ospedaliero Universitaria di Sassari, Sassari